CLINICAL TRIAL: NCT06784232
Title: Alveolar Ridge Preservation: Biologically-oriented Alveolar Ridge Preservation Vs Modified Periosteal Inhibition
Status: Active, not recruiting | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: PERIOSTEAL INHIBITION
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Ridge Preservation; Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — alveolar bone specimens withdrawn with trephine bur
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BARP: collagen-bonegraft-collagen
  Interventions: Procedure: BARP
- Modified Periosteal Inhibition Technique: cortical lamina, human fibrin glue and collagen
  Interventions: Procedure: Modified Periosteal Inhibition Technique

INTERVENTIONS:
Procedure: BARP — deep layers of collagen, medium-superficial heterologous bone graft, superficial collagen layer
  Groups: BARP
Procedure: Modified Periosteal Inhibition Technique — Cortical lamina stabilized with human fibrin glue to preserve the buccal wall of the socket. The socket was then filled with collagen.
  Groups: Modified Periosteal Inhibition Technique

SUMMARY:
The modified periosteal inhibition technique has been proposed as an alternative to limit crestal resorption following tooth extraction in sockets with a residual vestibular thickness of <1 mm. This technique aims to prevent osteolytic activity on the external surface of a post-extraction socket by applying a 0.5 mm-thick soft cortical plate of porcine origin, secured with fibrin glue. By avoiding the placement of bone graft material inside the socket, the technique seeks to effectively counteract bone remodeling, achieving minimal reduction in the size of the alveolar crest.

The aim is to evaluate the effectiveness of the modified periosteal inhibition technique in preserving the dimensions of the alveolar ridge after tooth extraction, by comparing it with the Biologically-oriented Alveolar Ridge Preservation technique.

DETAILED DESCRIPTION:
The primary objective of the study is to clinically compare the effect on the preservation of the alveolar ridge using the modified periosteal inhibition technique and the Biologically-oriented Alveolar Ridge Preservation technique.

The secondary objective is the collection of histological and histomorphometric data that allow to evaluate the quality and quantity of newly formed bone.

Study design: Observational study of a prospective non-profit cohort.

Study population: The study will be conducted in an outpatient hospital setting.

Number of patients to be enrolled to compare modified periosteal inhibition technique and BARP: 30 patients in the University of Trieste including dropouts.

Enrollment procedure: all patients who meet the inclusion and exclusion criteria will be enrolled in the study following the administration of the Information Sheet and the acquisition of informed consent.

The choice of the alveolar ridge preservation protocol will be motivated by the clinicians experience and the patients preference among those currently validated.

BARP: under local anesthesia, the compromised tooth will be extracted atraumatically without raising a flap. After granulation tissue removal, the socket will be filled with a collagen sponge (deep collagen layer) up to 4 to 5 mm from the most coronal extensions of the buccal crest to create a support for the intra-alveolar graft. A bovine derived xenograft will be placed on top of the collagen sponge to fill the coronal part of the socket, avoiding overfilling (graft layer). Socket sealing will be performed with a new layer of collagen sponge that will be placed over the exposed portion of the graft layer and firmly held by sutures.

Modified periosteal inhibition technique: under local anesthesia, an atraumatic tooth extraction will be performed, ensuring the preservation of the buccal bone. After granulation tissue removal, papillae incisions will be made, followed by an intra-sulcular incision along the buccal side of the socket, extending to the mesial and distal mid-tooth regions. A full-thickness flap will be elevated, creating sufficient space within the socket for the insertion of the cortical lamina. The lamina will be trimmed to the required shape, extending to the mesial and distal edges of the extraction socket. A few drops of human fibrin glue (2-3) will be applied to the cortical lamina, which will then be gently pressed against the buccal bone to secure it in place. A collagen sponge will be placed inside the socket to stabilize the clot and held in position with a suture.

For all patients, after 26 weeks of healing, a mucoperiosteal flap will be raised to expose the target site and a titanium implant will be inserted. During this phase, using a core drill to prepare the implant site, it will also be functional to obtain a bone sample that will be subsequently analyzed.

Study Outcomes

The primary endpoint is the width of the alveolar ridge, which will be assessed in two stages:

T0: initial condition of the alveolar ridge, measured before performing surgery; T1: final condition of the alveolar ridge, measured before implant insertion at 26 weeks of healing from surgery.

The primary endpoint will be classified as follows. The secondary endpoints are represented by histomorphometric variables: newly formed mineralized tissue (New bone/Total volume), graft residues (RG/TV), newly formed non-mineralized tissue (Nonmineralised tissue/Total volume), total mineralized tissue that will be assessed at twenty-six weeks of healing (Mineralised tissue/total volume) evaluated as means and standard deviations and with χ2 test.

The primary endpoint will then be assessed in relation to complications and adverse events, such as: soft tissue dehiscence; graft exposure; graft loss and wound infections.

The width of the alveolar ridge will be measured linearly and volumetrically, using digital scans processed by a 3D scanning software (Geomagic Control X, 3D System, Morrisville, USA) at the University of Trieste.

The data collected at follow-up and the outcome data are based on a clinical evaluation, considering the possible presence of complications and adverse events.

The histological and histomorphometric analysis of all samples will be performed by one of the authors, blinded to the study design and the origin of the biopsy. The biopsies, left inside the core drills to maintain the orientation of the bone core, will be rinsed with a cold 5% glucose solution to remove blood residues while maintaining the correct osmolarity (278 mOsm/L). The samples will then be fixed for 3 days in a 10% buffered formalin solution at pH 7.2 and then processed for histological and histomorphometric evaluation at the Bone Lab, University of Trieste. After this, the samples will be delivered to specialized and authorized companies for disposal, according to current legislation.

Collected data variables and sources The following variables will be collected for each enrolled patient/participant: width of the alveolar ridge; newly formed mineralized tissue; graft residues; non-mineralized newly formed tissue and total mineralized tissue.

Histological and histomorphometric analysis of all samples will be performed by one of the authors, blinded to the study design and biopsy origin. Biopsies, left inside the core drills to maintain the orientation of the bone core, will be rinsed with a cold 5% glucose solution to remove blood residues while maintaining the correct osmolarity (278 mOsm/L). Samples will then be fixed for 3 days in a 10% buffered formalin solution at pH 7.2 and then dehydrated in ascending series of alcohol rinses. After 5 days of preinfiltration in a 50% resin/alcohol solution, biopsies will be removed from the core drills and sample infiltration will be completed with methacrylate resin. After 12 days of polymerization, the samples will be cut along their longitudinal axis using a high-precision silicon carbide disc at 50 μm and then finished under running water with a series of polishing discs at approximately 30 ± 10 μm. They will then be mounted on slides and stained with acid fuchsin, toluidine blue and Von Kossa.

Following histological and histomorphometric analyses, the samples will be delivered to specialized and authorized companies for disposal, according to current legislation.

Statistical plan The statistical analysis will be performed by means of a computerized statistical package (SigmaStat 3.5, SPSS Inc., Germany). The data will be expressed as mean ± standard deviation and median (interquartile range), respectively, for parametric and non-parametric values.

Sample size calculation The aim of the study is to clinically compare different alveolar ridge preservation techniques. Considering the outcomes of previously published studies, it was calculated that will be necessary to recruit 15 patients for each group to obtain a statistically significant result through a comparison between subpopulations with a statistical power of 95% and a significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* Single-rooted tooth with indication for extraction with sockets having a residual thickness of <1 mm in the first 3 mm of the buccal residual crest presenting adjacent teeth;
* American Society of Anesthesiologists 3;
* Periodontal health or stability;
* Signature of informed consent.

Exclusion Criteria:

* Presence of periapical cystic lesions at the intervention sites;
* Loss of bone tissue extending to the apical third on radiographic examination;
* Extraction of adjacent teeth within a period ranging from 6 months prior to 6 months after the extraction;
* Lack of one or more walls of the post-extraction socket;
* Presence of general contraindications for oral surgery;
* Presence of inflammatory and autoimmune diseases;
* Uncontrolled diabetes (HbA1c 7%);
* History of tumors requiring chemotherapy or radiotherapy in the last 5 years;
* Previous therapy with bisphosphonates or high-dose corticosteroid therapy;
* Smoking (10 cigarettes/day);
* Allergy to bovine collagen;
* Pregnancy or breastfeeding;
* Lack of compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in an outpatient hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ridge width reduction | 26 weeks after tooth extraction and preservation tecnhique
  optical scanning comparison measured in millimetres at the mid-buccal and mid-palatal aspect of the socket
ridge height reduction | 26 weeks after tooth extraction and preservation tecnhique
  optical scanning comparison measured in millimetres at the mid-buccal, mid-palatal, mesial and distal aspect of the socket

SECONDARY OUTCOMES:
histologic and histomorphometric analysis of new bone formation | 26 weeks after tooth extraction and preservation tecnhique
  percentage of newly formed bone area to total measured area
histologic and histomorphometric analysis of residual graft particles | 26 weeks after tooth extraction and preservation tecnhique
  percentage of graft particles area to total measured area
histologic and histomorphometric analysis of marrow spaces | 26 weeks after tooth extraction and preservation tecnhique
  percentage of soft tissue area to total measured area

CONTACTS AND LOCATIONS:
Locations (1):
- University of Trieste, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No